CLINICAL TRIAL: NCT04037176
Title: Treatment With Omalizumab in Food Allergic Children (TOFAC)
Brief Title: Behandling af Boern Med Foedevareallergi Med Omalizumab (Xolair)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Carsten Bindslev-Jensen (Other)
Collaborators: Novartis Pharmaceuticals (Industry); Thermo Fisher Scientific, Inc (Industry)
Responsible Party: Sponsor-Investigator, Carsten Bindslev-Jensen, Professor, M.D., Dr.Med. Ph.D,, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EudraCT 2018-004427-37
Record Dates: First submitted 2019-05-10; First posted 2019-07-30 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Food Allergy
Keywords: Omalizumab; Xolair
MeSH Terms: conditions — Food Hypersensitivity | interventions — Omalizumab

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomized to treatment with Omalizumab (regular dose of asthma dosing according to total IgE and weight) or placebo (3:1). Primary endpoint after 3 months treatment.
  Responders (in the active as well as the placebo group) will continue treatment with the same dose of Omalizumab/placebo for a further 3 months. All non-responders will receive maximum dose of Omalizumab (according to weight, but not total IgE) for another 3 months.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The syringes are filled and masked with opaque material of unblinded personnel who do not have patient contact.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omalizumab (Active Comparator): Omalizumab is a sterile solution in a prefilled syring for subcutaneous injection. The syrings contains 75 mg or 150 mg omalizumab.
  75 patients will have Omalizumab in doses depending of body weight and IgE every 2. or 4. week for 6 month Omalizumab is administered subcutaneously
  Interventions: Drug: Omalizumab
- Placebo (Placebo Comparator): Placebo contains sodium chloride 0,9 % in a prefilled syring for subcutaneous injection.
  25 patients will have placebo depending of the body weight and IgE every 2. or 4. week in 3 month. They will subsequently get Omalizumab for 3 month if nonresponders.
  Placebo is administered subcutaneously
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Omalizumab — Subcutaneous administration every 2. week or every 4. week. Dose is depending of the patients weight and IgE
  Other Names: Xolair
  Arms: Omalizumab
Other: Placebo — Subcutaneous administration every 2. week or every 4. week. Dose is depending of the patients weight and IgE
  Other Names: NaCl
  Arms: Placebo

SUMMARY:
Food allergy is a common disease in childhood affecting up to 8% of children in Westernized countries. About 30 percent of children with food allergies are allergic to more than one food, most often milk, egg, wheat, peanut and tree nut. Peanut and hazelnut are common triggers of severe and potentially fatal food-induced anaphylactic reactions. Currently, there is no curative treatment for food allergy. Novel therapies for this potentially life-threatening condition are therefore much needed.

DETAILED DESCRIPTION:
Randomized, double-blind, placebo-controlled study to study the effect of Omalizumab on children with food allergy.

Primary endpoint: Change in challenge threshold after 3 months of treatment in patients treated with Omalizumab versus placebo.

Secondary endpoints: Change in challenge threshold at 6 months. Change in Skin Prick Test (SPT), serum markers for allergy (specific IgE, IgG4, BAT (basofil activation test)), severity of comorbidity, and quality of life from at 3 and 6 months. Change in treshold within and between the groups.

The investigator's hypothesis is that increased Omalizumab dose and/or a longer treatment period will increase food allergy threshold.

Within the groups:

* 3 months treatment with Omalizumab in asthma dose versus 6 months with Omalizumab in asthma dose - in primary responders
* 3 months treatment with Omalizumab in asthma dosing versus 3 months additional treatment with Omalizumab in max dose - in primary non-responders
* 3 months treatment with placebo versus 6 months with placebo- in primary placebo-responders
* 3 months treatment with placebo versus 3 months with max dose Omalizumab - placebo cross over to active.

Between the groups:

* 3 months treatment with Omalizumab in asthma dose versus 3 months with max dose Omalizumab
* 6 months treatment with Omalizumab in asthma dose versus 3 months with max dose Omalizumab.

Patients are randomized electronically via an e-CRF prepared by OPEN in RedCap. Assigned 3:1 to Omalizumab or placebo in 13 x 8 block (6:2) by a blinded health care person.

GCP-monitoring is performed by the local GCP-unit at Odense University Hospital

ELIGIBILITY:
Inclusion Criteria:

* children between 6 and 18 years
* a clinical diagnosis of food allergy to ≥1 food allergen
* a positive SPT (mean wheal diameter > 3 mm)
* s-IgE > 0.35 kIU/l
* a positive food challenge with a threshold at or below 300 mg of protein (443 mg cumulative) in a double blind placebo controlled food challenge (DBPCFC).
* (If the patient is allergic to more than one food allergen, the allergen with the highest probability of fulfilling the inclusion criteria (based on case history, level of s-IgE and when available challenge results within the last year) will be used).

Exclusion Criteria:

* t-IgE >1500 kIU/L.
* Significant co-morbidity that might compromise the patient's safety or study outcomes.
* Pregnancy or nursing in the adolescents. Women of childbearing potential have to use safe contraception (intrauterine device or hormonal contraception if sexual active). Safe contraception has to be used during the whole trial period and half a year after the last dose of the trial medicine has been taken.
* Ongoing treatment with antihistamine or drugs with antihistaminic properties that cannot be paused during the study
* Ongoing treatment with drugs that may impair safety during food challenge e.g. β-blockers or ACE-inhibitors that cannot be paused during the study
* Ongoing treatment with oral glucocorticoids/Omalizumab/allergen immunotherapy (AIT)
* Alcohol abuse, abuse of opioids or other drugs in adolescents
* Treated with Omalizumab until ½ years before the study
* Patients/parents who are not supposed to be able to meet the requirements in the protocol
* Patients/parents who are physically or mentally unable to consent
* Patients who have reduced liver function or kidney function

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Change in challenge threshold (mg food protein tolerated by oral intake) | 0-3 months
  Change in challenge threshold after 3 months of treatment in patients treated with Omalizumab versus placebo

SECONDARY OUTCOMES:
Change in quality of life (validated questionnaire - food allergy quality of life questionnaire (FAQLQ)) | 0-6 months
  To estimate improvement in QoL before and after 3 months and 6 months treatment, using FAQLQ on a seven point scale with one as the best possible score (score 1-7)
Change in skin prick test size (mm) | 0-6 months
  To estimate changes in skin prick test size during the treatment
Change in severity of co-morbidity (atopic dermatitis, asthma, allergic rhintitis using clinical severity scores) | 0-6 months
  To estimate improvement in atopic diseases by evaluation of disease severity (SCORAD atopic dermatitis, VAS and CSMS rhinitis, ATC asthma)
Change in levels of serum markers for food allergy (IgE (kIU/L), IgG4 (kIU)) | 0-6 months
  To estimate changes in serum markers for allergy during the treatment
Change in levels of serum markers for food allergy BAT test (CD-sens)) | 0-6 months
  To estimate changes in serum markers for allergy during the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Bindslev-Jensen, Prof DM PhD, Study Director — Odense Research Center For Anaphylaxis; Susanne Halken, Prof DM MD, Study Chair — Department of Childrens Hospital
Locations (1):
- Odense Research Center for Anaphylaxis, Allergy Center, Odense University Hospital, Odense C, Funen, Denmark